CLINICAL TRIAL: NCT01048307
Title: Randomised, Controlled, Clinical Trial on the Safety and Efficacy of Prontosan Wound Irrigation Solution Compared to Standard Therapy in the Treatment of Hard-to-Heal Venous Leg Ulcers
Brief Title: Effect of Prontosan Wound Irrigation Solution on Venous Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Calvary Hospital, Bronx, NY (Other)
Collaborators: B. Braun Medical SA (Industry)
Responsible Party: Ali Koca, MD, B. Braun Medical Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPM-I-H-0902
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Wound Care; Venous Ulcer Care; Wound Cleansing; Chronic Wound Care
Keywords: prontosan; wound cleansing; wound irrigation; phmb; polihexanide; betaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prontosan wound irrigation solution (Experimental): Prontosan® Wound Irrigation Solution (experimental group):
  * cleansing the wound bed at dressing change with Prontosan® Wound Irrigation Solution; a sterile gauze dressing impregnated with the Prontosan® solution will be placed on the wound in the form of a moist compress and removed after approx.15 minutes;
  * placing the primary dressing (Profore® WCL): the dressing will be impregnated with Prontosan® Wound Irrigation Solution;
  * fixing the dressing to the wound using multilayered elastic compression bandaging (Profore®bandaging system).
  Interventions: Device: Prontosan wound irrigation solution
- Saline irrigation (standard care control) (Placebo Comparator): Saline (control group):
  * cleansing the wound bed at dressing change with saline; a sterile gauze dressing impregnated with the saline will be placed on the wound in the form of a moist compress and removed after approx.15 minutes;
  * placing the primary dressing (Profore® WCL): the dressing will be impregnated with saline;
  * fixing the dressing to the wound using multilayered elastic compression bandaging (Profore® bandaging system).
  Interventions: Device: Prontosan wound irrigation solution

INTERVENTIONS:
Device: Prontosan wound irrigation solution — Prontosan® Wound Irrigation Solution (experimental group):
  • Active ingredients (Polihexanide 0.1%, Betaine 0.1%) cleansing the wound bed at dressing change with Prontosan® Wound
  Saline (control group):
  * cleansing the wound bed at dressing change with saline; a sterile gauze dressing impregnated with the saline will be placed on the wound in the form of a moist compress and removed after approx.15 minutes;
  * placing the primary dressing (Profore® WCL): the dressing will be impregnated with saline;
  * fixing the dressing to the wound using multilayered elastic compression bandaging (Profore® bandaging system).
  Other Names: Wound irrigation solution containing PHMB; Polihexanide; Betaine; Wound cleanser

SUMMARY:
Objective:

To evaluate the efficacy and safety of Prontosan® Wound Irrigation Solution in the treatment of hard-to-heal venous leg ulcers compared to wound irrigation with saline solution

Methodology:

Randomised, controlled multi-centre, prospective clinical trial

Planned number of subjects:

20 patients in experimental group (Prontosan® Wound Irrigation Solution) 8 patients in control group (wound irrigation with saline)

Products under investigation:

Prontosan® Wound Irrigation Solution

Study Duration:

3-4 weeks

DETAILED DESCRIPTION:
Investigational product, dose and administration:

Prontosan® Wound Irrigation Solution (experimental group) and saline solution (control group) will be applied at inclusion and reapplied after dressing changes.

The treatment scheme is as follows:

1. Prontosan® Wound Irrigation Solution (experimental group):

   * cleansing the wound bed at dressing change with Prontosan® Wound Irrigation Solution; a sterile gauze dressing impregnated with the Prontosan® solution will be placed on the immediate wound in the form of a moist compress and removed after approximately 15 minutes;
   * placing the primary dressing (Profore® WCL): the dressing will be impregnated with Prontosan® Wound Irrigation Solution;
   * fixing the dressing to the wound using multilayered elastic compression bandaging (Profore® bandaging system).
2. Saline (control group):

   * cleansing the wound bed at dressing change with saline; a sterile gauze dressing impregnated with the saline will be placed on the wound in the form of a moist compress and removed after approx.15 minutes;
   * placing the primary dressing (Profore® WCL): the dressing will be impregnated with saline;
   * fixing the dressing to the wound using multilayered elastic compression bandaging (Profore® bandaging system).

Dressings will be changed and the treatment procedure will be repeated in the clinic 2x/weekly or more. The efficacy of the treatment procedure will be evaluated on the basis of a 2 week observation period.

Treatment efficacy assessment:

* Assessment of clinical signs and symptoms at entry to the study and after one and two weeks.
* Quantitative and qualitative microbiological analysis at entry to the study and after two weeks.
* Wound planimetry using PictZar® CDM at entry to the study and after two weeks.

Primary aim:

* clinical signs assessed by:

  1. reduction of slough and necrotic tissue
  2. control of exudate
  3. presence of granulation tissue
* reduction of inflammatory signs (surrounding skin)
* reduction in wound size (assessed by wound planimetry)
* reduction of bacterial load (quantitative and qualitative microbiological

Secondary aim:

- tolerance and safety assessment:

1. adverse drug reaction
2. adverse events
3. early withdrawal from the study

ELIGIBILITY:
Inclusion Criteria:

* males and females aged at least 18 with wounds of venous aetiology (documented by targeted exams) located in the lower limbs
* Ankle Brachial Index (ABI) ≥ 0.7
* patients who have not had an antimicrobial (systemic antibiotic or topical antiseptic) over the 30 days before joining the study

Exclusion Criteria:

Exclusion criteria

* age below 18 years
* presence of clinical infection, or current use of antiseptics or antibiotics
* chronic wounds of long duration (>30cm2 and >1 year duration)
* involvement in other wound related trials within the past 30 days
* sensitivity to any of the components of Prontosan® or dressing material
* intolerance to compression therapy
* active osteomyelitis in the ulceration area
* active rheumatoid arthritis (RA) requiring any immunosuppressive therapy
* collagen vascular disease active treated with steroids
* chronic diseases that could impact the course of the study (malicious cancer, TB, AIDS, mental illnesses)
* plasma protein below 4 g/dl
* anaemia: haemoglobin below 10 g/dl
* both, controlled and uncontrolled diabetics (type 1 or 2)
* patients on any rheological agents (not including aspirin)

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Reduction of bacterial burden (quantitative bacteriology) Reduction in slough and necrotic tissue (clinical score) Amount and quality of granulation tissue (clinical score) Exudate type and amount (clinical score) | weekly

SECONDARY OUTCOMES:
Adverse device effect (s) Adverse events | volunteered at any time or during weekly evaluation visits

CONTACTS AND LOCATIONS:
Overall Officials: Oscar M Alvarez, PhD, Principal Investigator — Calvary Hospital, Wound Care; Martin Wendelken, RN, DPM, Study Director — Calvary Hospital, Wound Care
Locations (1):
- Calvary hospital center for curative and palliative wound care, The Bronx, New York, United States